CLINICAL TRIAL: NCT07298681
Title: The Effect of Benner's Jigsaw Teaching Technique Based on the Novice to Expert Model and Scenario-Based Peripheral Intravenous Catheterization Instruction on Skill Acquisition of Nursing Students: An Experimental Study.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Ayşe ULUÇAY HAMARAT, Sub-ınvestigator, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Cumhuriyet University Nursing; 2025-10/37 (Other: Sivas Cumhuriyet Üniversitesi Sağlık Bilimleri Araştırmaları Etik Kurulu)
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Nursing Education; Clinical Skills Training
Keywords: Jigsaw Teaching Method; Scenario-Based Learning; Skill Acquisition; Nursing Students; Educational Intervention

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either the intervention group or the control group in a parallel design to compare the effects of a structured educational approach on clinical skill performance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jigsaw and Scenario-Based Training (Experimental): Participants in this arm will receive training on peripheral intravenous catheter (PIVC) insertion using the Jigsaw cooperative learning method combined with scenario-based education. The training includes group-based learning, structured scenarios, skill demonstration, and supervised practice.
  Interventions: Behavioral: Jigsaw and Scenario-Based Training
- Traditional Training (Active Comparator): Participants in this arm will receive traditional/standard training for peripheral intravenous catheter (PIVC) insertion, including lecture-based instruction, demonstration, and supervised skills practice without Jigsaw or scenario-based components.
  Interventions: Behavioral: Traditional Training

INTERVENTIONS:
Behavioral: Jigsaw and Scenario-Based Training — A structured educational program combining the Jigsaw cooperative learning method with scenario-based training to improve peripheral intravenous catheter (PIVC) insertion skills. Training includes group-based learning, scenario discussions, skill demonstration, and supervised practice.
  Arms: Jigsaw and Scenario-Based Training
Behavioral: Traditional Training — Standard instructional approach including lecture-based teaching, demonstration, and supervised practice for peripheral intravenous catheter (PIVC) insertion, without Jigsaw or scenario-based components.
  Arms: Traditional Training

SUMMARY:
This randomized controlled experimental study aims to evaluate the effectiveness of a training program based on the Jigsaw teaching technique and scenario-based learning in improving the peripheral intravenous catheterization skill levels of first-year nursing students. Participants will be randomly assigned to either the intervention group, receiving Jigsaw-based collaborative learning combined with clinical scenarios, or the control group receiving traditional skills training. The primary outcome is the improvement in students' clinical skill performance as measured by a standardized skill assessment checklist. The study seeks to determine whether innovative, active learning methods can enhance fundamental nursing skills training

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of a structured educational intervention based on the Jigsaw teaching technique combined with scenario-based clinical training on the skill performance of first-year nursing students. The study is designed as a randomized controlled experimental trial.

The intervention group will receive a structured education program that includes collaborative learning through the Jigsaw method, scenario-based skill practice, and guided feedback. The control group will receive standard skills laboratory training provided within the regular curriculum. All students will complete the same skill performance assessment before and after the intervention.

The primary objective of the study is to determine whether the combined Jigsaw and scenario-based educational approach improves students' practical skill performance compared to standard training. Secondary objectives include evaluating changes in students' self-confidence, engagement in the learning process, and satisfaction with the educational method.

The study will be conducted in a controlled laboratory environment, and all participants will be randomly assigned to the intervention or control group. The results are expected to contribute to the development of innovative and effective teaching strategies for fundamental nursing skills education.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research
* To be a first-year Nursing student
* To be taking the Nursing Fundamentals-II course for the first time
* To be a smart phone or computerVolunteering to participate in resrs a day

Exclusion Criteria:

* Being a foreign national (due to the risk of having language problems)
* To have received high school and associate degree education in the field of Public health

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Peripheral Intravenous Catheter (PIVC) Insertion Skill Score | Immediately post-intervention
  Change in students' PIVC insertion skill performance measured using a standardized skill checklist. Scores will be obtained immediately after the training intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Şerife KARAGÖZOĞLU, PhD, Professor, Study Chair — Cumhuriyet University
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No